CLINICAL TRIAL: NCT04062916
Title: Improvement in Quality of Life and Pain Scores After Laparoscopic Management of Deep Infiltrating Endometriosis
Status: Completed | Type: Observational
Sponsor: Acibadem Fulya Hastanesi (Network)
Responsible Party: Sponsor
Other Study IDs: AcibademFulyaHendo
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Endometriosis
Keywords: endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women with endometriosis: 65 women whose main symptom was pain and who did not respond to medical treatment and underwent endometriosis surgery
  Interventions: Other: BSGE pelvic pain questionnaire and VAS scores

INTERVENTIONS:
Other: BSGE pelvic pain questionnaire and VAS scores — Patients were evaluated using the BSGE pelvic pain questionnaire in terms of pre-operative and post-operative pain assessment in order to determine the effects of endometriosis surgery on the quality of life. The patients were asked to indicate their levels of dyspareunia, dysmenorrhea, and chronic pelvic pain on a VAS on the pelvic pain questionnaire.

SUMMARY:
This is a retrospective cohort study that evaluates the postoperative pain findings of a consecutive series of laparoscopic surgeries for deep infiltrating endometriosis (DIE).

DETAILED DESCRIPTION:
The study was carried out in university hospitals (Istanbul, Turkey). Patients diagnosed through bimanual gynecologic examination, gynecologic ultrasound or magnetic resonance imaging-confirmed endometrioma and DIE together; who underwent a laparoscopic surgery by a team of gynecologists, colorectal surgeons, and a urologist were retrospectively evaluated. The data were collected in a specific database and analyzed for postoperative pain outcomes through a comparison with preoperative symptoms scored using a visual analogue score (VAS), and the British Society of Gynecologic Endoscopy (BSGE) pelvic pain questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with deep infiltration endometriosis and endometrioma diagnosed through bimanual gynecologic examination, gynecologic ultrasound or through laparoscopically confirmed endometrioma and DIE together;
* DIE with bowel involvement that required shaving or segmental resection for colorectal lesions and nodules;
* Who completed the VAS score and BSGE questionnaire;
* Follow-up period of at least 3 months;
* Patients resistant to medical therapy (NSAIDs, OCPs, levonorgestrel-releasing intrauterine device (IUD), and progesterone) or refuse to use medical therapy.

Exclusion Criteria:

*Any other endometriosis patient that do no meet the inclusion criteria

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with endometriosis 65 women whose main symptom was pain and who did not respond to medical treatment and underwent endometriosis surgery
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life after endometriosis surgery | 7 years
  Effects of endometriosis surgery on the quality of life by using BSGE pelvic pain questionnaire
Pain levels after endometriosis surgery | 3 years
  Effects of endometriosis surgery on pelvic pain by using VAS scores

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Bastu, MSc, MD, Principal Investigator — Acibadem Fulya Hospital
Locations (1):
- Acibadem Fulya Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided